CLINICAL TRIAL: NCT05207618
Title: Utility of the Administration of Tannin Specific Natural Extract, Chesnut and Quebracho Based, for Irritable Bowel Syndrome Diarrhea Predominant
Brief Title: Utility of the Administration of Chesnut and Quebracho Extract for Irritable Bowel Syndrome Diarrhea Predominant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas José de San Martín (Other)
Collaborators: SILVATEAM (Unknown)
Responsible Party: Principal Investigator, Maria Marta Piskorz, Neurogastroenterologist at Hospital de Clinicas, Principal Investigator, Hospital de Clinicas José de San Martín
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25130271
Record Dates: First submitted 2021-12-09; First posted 2022-01-26 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Irritable Bowel Syndrome; Diarrhea
Keywords: intestinal microbiota; intestinal permeability; intestinal inflammation
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea

STUDY DESIGN:
Intervention Model Description: before- after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBS PATIENTS (Experimental): Natural specific tannin, chestnut
  Interventions: Dietary Supplement: ARBOX (QUEBRACHO AND CHESNUT EXTRACT)

INTERVENTIONS:
Dietary Supplement: ARBOX (QUEBRACHO AND CHESNUT EXTRACT) — ARBOX TWICE A DAY FOR 60 days

SUMMARY:
Irritable bowel syndrome is a highly prevalent disorder and consumes many health resources. Its physiopathogenesis is multifactorial. Some of the factors involved have to do with the alteration of the intestinal microbiota, low-grade inflammation and the alteration of intestinal permeability. Specific tannins have been shown to have prebiotic effects and could be useful in treating this condition. This is an exploratory before-after study that aims to evaluate the effect of a chestnut and quebracho extract on the symptoms of IBS diarrhea predominant, serum cytokine levels, microbiota and intestinal permeability, as well as on metabolomics.

DETAILED DESCRIPTION:
In vitro studies have shown that chestnut and quebracho extract has a prebiotic effect of modulating the intestinal microbiota, but also, bacterial fermentation produces metabolites with powerful anti-inflammatory effects such as quecetin. Irritable bowel syndrome (IBS) is a multifactorial disorder involving factors related to the intestinal microbiota, low-grade inflammation, and impaired intestinal permeability.

In this study, 30 patients with predominant IBS diarrhea and 50 healthy controls will be included. IBS patients will receive chestnut and quebracho extract twice a day for 8 weeks. They will be measured at baseline and at 8 weeks: 27 serum pro and anti-inflammatory cytokines and serum zonulin. Likewise, the intestinal microbiota and metabolomics will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* IBS patients: Both sexes with a diagnosis of irritable bowel syndrome variety diarrhea according to the Rome IV criteria

Healthy Controls: Relatives of patients who do not show any disease, who do not take medication or present symptoms.

Exclusion Criteria:

* patients with digestive tract disease,
* systemic diseases such as severe heart, kidney or liver failure,
* history of previously known digestive tract surgeries and / or intestinal adhesions,
* diabetes mellitus,
* cirrhosis,
* inflammatory bowel disease,
* celiac disease,
* patients with cognitive impairment,
* alcoholics,
* lack of consent .
* patients who have received antibiotics in the last month.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Change in Irritable bowel syndrome symptoms severity (IBS severity score, 75-500) | 60 days
  Change in IBS severity score from baseline
Change in Stool frequency (number of deposition per day) | 60 days
  Change in stool frequency per day from baseline
Change in Stool consistency (Bristol stool form scale, 1-7) | 60 days
  Change in Stool consistency from baseline

SECONDARY OUTCOMES:
Change in Inflammation | 60 days
  serum cytokine level change from baseline. Bioplex Biorad
Change in Intestinal permeability | 60 days
  Change in Anti Zonuline level from baseline
Change in Intestinal microbiota | 60 days
  change in 16-s sequency from baseline

CONTACTS AND LOCATIONS:
Overall Officials: MARIA MARTA PISKORZ, Principal Investigator — NEUROGASTROENTEROLOGIA HOSPITAL DE CLINICAS
Locations (1):
- Hospital de Clinicas Jose de San Martin. Buenos Aires University, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No